CLINICAL TRIAL: NCT00116896
Title: Phase I Study of OSI-7904L in Combination With Cisplatin in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of Cisplatin Plus OSI-7904L in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: OSI-904-102
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2003-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — ((S)-2-(5-(1,2-dihydro-3-methyl-1-oxobenzo(f)-quinazoline-9-yl)methyl)amino-1-oxo-2-isoindolynyl)-glutaric acid; Cisplatin

INTERVENTIONS:
Drug: OSI-7904L
Drug: Cisplatin

SUMMARY:
This is a Phase I, open-label, dose escalation, study of the combination of cisplatin and OSI-7904L given on Day 1 every 21 days in patient who have advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Advanced and/or metastatic solid tumor for which no effective therapy is available
* ECOG performance status 0-2
* Adequate bone marrow, hepatic and renal function

Exclusion Criteria:

* Patients with active or uncontrolled infections
* Neurotoxicity >= Grade 2
* Symptomatic brain metastases which are not stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-06; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Vanderbilt Universtiy Medical Center, Nashville, Tennessee
  - Institute for Drug DevelopmentCancer Therapy & Research Center, San Antonio, Texas